CLINICAL TRIAL: NCT04440709
Title: Restoration of Bimanual Activities of Daily Living Using a Brain/Neural Hand Exoskeleton (B/NHE) in Hand Paralysis
Brief Title: Brain/Neural Hand Exoskeleton Control for Restoration of Bimanual Tasks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Charite University, Berlin, Germany (Other); Reutlingen University (Unknown); Hochschule der Medien (Unknown); University of Stuttgart (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NEU007/1
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injury; Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain/neural hand exoskeleton (B/NHE) (Experimental)
  Interventions: Device: Brain/neural hand exoskeleton (B/NHE)

INTERVENTIONS:
Device: Brain/neural hand exoskeleton (B/NHE) — The brain/neural hand exoskeleton restores hand motor function by translating user's intention into grasping motions

SUMMARY:
This study investigates whether spinal cord injury and stroke survivors (n=10) are able to operate a brain/neural hand exoskeleton (B/NHE) based on electroencephalography (EEG) and electrooculography (EOG) for restoration of bimanual activities of daily living (ADLs). To assess bimanual ADLs, the Berlin Bimanual Task Assessment (BEBITA) will be applied. Improvements in BEBITA will be evaluated with and without B/NHE use.

ELIGIBILITY:
Inclusion Criteria (Stroke):

* single ischemic or hemorrhagic insult with subcortical lesion (medullary canal, internal capsula, pedunculi cerebri)
* interval since stroke at least 6 months
* substantial motor deficit with:
* Medical Research Council (MRC) -score of less than 2 out of 6 possible points (0=no activity; 1=visible contraction without motor effect; 2=movements with elimination of gravity; 3=movements against gravity; 4=movements against weak resistance; 5=normal force)
* Fugl-Meyer Test (upper extremity) of less than 31 points, "no to little mobility"

Inclusion Criteria (Spinal Cord Injury):

* cervical spinal cord injury, height C5-C6
* interval after spinal cord injury at least 6 months
* substantial motor deficit with American Spinal Cord Association (ASIA) -Classification B or C (A=no muscle function/sensitivity below the spinal cord injury; B=no muscle function, limited sensitivity present; C=low non-relevant muscle function, sensitivity present; D=functionally relevant muscle functions present; E=fully preserved or restored functions)

Exclusion Criteria (Stroke and Spinal Cord Injury):

* Alcohol or drug problem (regular consumption of more than 2 alcoholic beverages per day, or taking illegal drugs)
* currently undergoing neurological or psychiatric treatment based on a secondary diagnosis
* Severe and uncontrollable medical problems:
* Non-adjusted malignant high blood pressure, World Health Organization (WHO) Hypertension Grade II
* non-adjustable diabetes mellitus, HbA1c > 58 mmol/mol
* renal failure, from KDIGO glomerular filtration rate (GFR) category G3b (moderate to severe impairment)
* Liver failure, Child-Pugh stages B and C
* Heart failure New York Heart Association (NYHA) grade III-IV
* malignant tumor disease
* severe arrhythmia in need of treatment
* severe oedemas
* severe arthritis
* serious cognitive impairment (minimum status below 23 points)
* Severe spasticity (Ashworth grade ≥ 4)
* Pregnancy
* Bilateral motor deficit (in stroke patients)

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in Berlin Bimanual Task Assessment (BEBITA) score | Hand function will be assessed twice on the same day. Once before the hand exoskeleton is applied (absence of the assistive device) and once after the brain-controlled hand exoskeleton was attached to the patients' hand and arm.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Charité - University Medicine Berlin, Berlin

REFERENCES:
- [Derived] Vermehren M, Colucci A, Angerhofer C, Peekhaus N, Kim WS, Chang WK, Kim H, Homberg V, Paik NJ, Soekadar SR. The Berlin bimanual test for stroke survivors (BeBiT-S): evaluating exoskeleton-assisted bimanual motor function after stroke. J Neuroeng Rehabil. 2025 Dec 8;22(1):261. doi: 10.1186/s12984-025-01822-6. PMID 41361479